CLINICAL TRIAL: NCT00337727
Title: A Randomized, Double-Blind, Parallel-Group Study Conducted Under In-House Blinding Conditions to Determine the Efficacy and Tolerability of Aprepitant for the Prevention of Chemotherapy Induced Nausea and Vomiting (CINV) Associated With Moderately Emetogenic Chemotherapy (MEC)
Brief Title: Aprepitant for the Prevention of Chemotherapy Induced Nausea and Vomiting (CINV)(0869-130)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0869-130; 2006_016 (Other: protocol number)
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2009-11-06 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Other): Arm 1: Day 1: aprepitant 125 mg capsule; ondansetron 8 mg capsule prior to chemotherapy and 1 8mg capsule 12 hrs after first dose; dexamethasone 12 mg tablets + 2 dexamethasone Pbo tablets. Day 2: Aprepitant 80 mg capsule; Ondansetron 8 mg capsule every 12 hours Day 3: Aprepitant 80 mg capsule Ondansetron 8 mg capsule every 12 hours.
  Interventions: Drug: aprepitant; Drug: Comparator: ondansetron; Drug: Comparator: dexamethasone; Drug: Comparator; Placebo (unspecified)
- 2 (Other): Arm 2: Day 1: Aprepitant 125 mg Pbo capsule; Ondansetron 8 mg capsule prior to chemotherapy and 8 mg capsule 12 hours after first dose; Dexamethasone 20 mg tablets. Day 2: Aprepitant 80 mg Pbo capsule; Ondansetron 8 mg capsule every 12 hours; Day 3: Aprepitant 80 mg Pbo capsule; Ondansetron 8 mg capsule every 12 hours. 3 Day treatment period Optional cycle 2 is being offered to patients. Optional cycle 2 will substitute aprepitant with fosaprepitant dimeglumine 115 mg or Pbo on day 1. All other dosing regimen will remain the same as cycle 1.
  Interventions: Drug: Comparator: ondansetron; Drug: Comparator: dexamethasone; Drug: Comparator: fosaprepitant dimeglumine; Drug: Comparator; Placebo (unspecified)

INTERVENTIONS:
Drug: aprepitant — aprepitant 125 mg capsule; aprepitant 80 mg capsule Three day treatment period.
  Other Names: MK0869
  Arms: 1
Drug: Comparator: ondansetron — Ondansetron 8 mg capsule Three day treatment period.
  Other Names: Zofran®
Drug: Comparator: dexamethasone — dexamethasone 12 mg tablets; 20 mg tablets Three day treatment period.
  Other Names: DEXAMETHASONE TABLETS USP
Drug: Comparator: fosaprepitant dimeglumine — fosaprepitant dimeglumine 115 mg
  Other Names: EMEND®
  Arms: 2
Drug: Comparator; Placebo (unspecified) — dexamethasone 12mg Pbo tablets.
  Arms: 1
Drug: Comparator; Placebo (unspecified) — Aprepitant 80 mg & 125 mg Pbo capsules.
  Arms: 2

SUMMARY:
The study will test aprepitant for the prevention of CINV in patients receiving their initial cycle of Moderately Emetogenic Chemotherapy (MEC). Patients receiving more then one cycle of chemotherapy may opt to participate in an optional second cycle during which the patient will receive the same antiemetic regimen as cycle 1, except that an IV formulation of aprepitant will be given in place of the oral formulation on study day one. Study drug administration on subsequent days will be given orally as in cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be naive to emetogenic chemotherapy with histologically or cytologically confirmed malignant disease scheduled to receive a single dose of moderately emetogenic chemotherapy on study day 1
* Karnofsky score of 60 or greater

Exclusion Criteria:

* Patient is scheduled to receive any dose of cisplatin
* Patient will receive abdominal or pelvic radiation a week prior and up to 6 days after initiation of chemotherapy
* Any allergies to study drug or antiemetics
* Taking CYP3A4 substrates/prohibited medication
* Significant medical or mental conditions
* Abnormal laboratory values (platelets, absolute neutrophils, AST, ALT, bilirubin or creatinine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2008-10-28 (Actual); Study Completion 2008-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rapoport BL, Jordan K, Boice JA, Taylor A, Brown C, Hardwick JS, Carides A, Webb T, Schmoll HJ. Aprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with a broad range of moderately emetogenic chemotherapies and tumor types: a randomized, double-blind study. Support Care Cancer. 2010 Apr;18(4):423-31. doi: 10.1007/s00520-009-0680-9. Epub 2009 Jul 1. PMID 19568773
- [Derived] Rapoport BL. Efficacy of a triple antiemetic regimen with aprepitant for the prevention of chemotherapy-induced nausea and vomiting: effects of gender, age, and region. Curr Med Res Opin. 2014 Sep;30(9):1875-81. doi: 10.1185/03007995.2014.925866. Epub 2014 Jun 12. PMID 24911369
- [Derived] Aapro MS, Schmoll HJ, Jahn F, Carides AD, Webb RT. Review of the efficacy of aprepitant for the prevention of chemotherapy-induced nausea and vomiting in a range of tumor types. Cancer Treat Rev. 2013 Feb;39(1):113-7. doi: 10.1016/j.ctrv.2012.09.002. Epub 2012 Oct 11. PMID 23062719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 58 investigative sites worldwide. The first patient entered the study on 16-Jan-
  2007 and the last patient's last visit was on 28-Oct-2008.
Pre-assignment Details: Cancer patients naïve to both moderately and highly emetogenic chemotherapy (MEC and HEC, respectively) scheduled to receive an initial course of MEC for confirmed malignant disease. The study focused on patients receiving an initial cycle of MEC (Cycle 1).
Groups:
- Aprepitant Regimen: Aprepitant 125mg by mouth (PO) plus ondansetron 8mg PO twice daily and dexamethasone 12mg PO on Day 1 and aprepitant 80mg PO once daily on Days 2 and 3.
- Standard Regimen: Ondansetron 8mg PO twice daily plus dexamethasone 20mg PO on Day 1 and ondansetron 8mg PO twice daily on Days 2 and 3.
Period: Overall Study
Arm/Group | Aprepitant Regimen | Standard Regimen
Started | 430 | 418
Completed | 412 | 406
Not Completed | 18 | 12
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 5 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant Regimen | Standard Regimen | Total
Number analyzed (Participants) | 430 | 418 | 848
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.8) | 55.9 (12.6) | 56.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 325 | 652
  Male | 103 | 93 | 196
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 287 | 296 | 583
  Asian | 49 | 35 | 84
  Black | 26 | 20 | 46
  Multi-racial | 50 | 53 | 103
  Other | 18 | 14 | 32
History of Motion Sickness [Number; unit: Participants]
  Yes | 24 | 41 | 65
  No | 405 | 376 | 781
  No Data - Assessment Not Completed | 1 | 1 | 2
History of Vomiting with Pregnancy [Number; unit: Participants] — Measure is specific to the female study population.
  Participants
    Yes | 61 | 75 | 136
    No | 266 | 250 | 516
    Not Applicable- Male Patients | 103 | 93 | 196

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Reported No Vomiting
Description: The number of patients who reported No Vomiting in the overall phase in Cycle
  1
Time Frame: Overall phase (0-120 hours post initiation of MEC) in Cycle 1.
Population: FAS (full analysis set) patient population was used for all efficacy evaluations and included patients who (1) received Moderately Emetogenic Chemotherapy (MEC), (2) took a dose of study drug, and (3) completed at least one post treatment efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Aprepitant Regimen | Standard Regimen
Number analyzed (Participants) | 425 | 406
Participants | 324 | 252
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Standard Regimen; Test type: Superiority or Other; p < 0.01, Regression, Logistic — Superiority based on 2-sided level of significance of 0.05, based on a logistic regression model that included terms for treatment group, region and gender

2. Secondary Outcome: Number of Patients Who Reported Complete Response
Description: The number of patients who reported Complete Response (no vomiting and no use of rescue medication) in the overall phase in Cycle 1.
Time Frame: Overall phase (0-120 hours post initiation of MEC) in Cycle 1
Population: FAS (full analysis set) patient population was used for all efficacy evaluations and included patients who (1) received MEC, (2) took a dose of study drug, and (3) completed at least one post treatment efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Aprepitant Regimen | Standard Regimen
Number analyzed (Participants) | 425 | 407
Participants | 292 | 229
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Standard Regimen; Test type: Superiority or Other; p < 0.01, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Aprepitant Regimen | Standard Regimen
Serious Adverse Events (participants affected / at risk) | 12/430 | 20/418
Other Adverse Events (participants affected / at risk) | 265/430 | 270/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant Regimen (N=430) | Standard Regimen (N=418)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial Occlusive Disease (Vascular disorders) | 0 | 1
Peripheral Ischemia (Vascular disorders) | 1 | 0
Superior Vena Cava Occlusion (Vascular disorders) | 1 | 0 — Superior Vena Cava Occlusion
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant Regimen (N=430) | Standard Regimen (N=418)
Neutropenia (Blood and lymphatic system disorders) | 10 | 9
Abdominal Pain (Gastrointestinal disorders) | 17 | 16
Abdominal Pain Upper (Gastrointestinal disorders) | 9 | 8
Constipation (Gastrointestinal disorders) | 37 | 53
Diarrhoea (Gastrointestinal disorders) | 40 | 46
Dyspepsia (Gastrointestinal disorders) | 14 | 13
Nausea (Gastrointestinal disorders) | 18 | 11
Vomiting (Gastrointestinal disorders) | 9 | 6
Asthenia (General disorders) | 26 | 23
Fatigue (General disorders) | 47 | 41
Mucosal Inflammation (General disorders) | 8 | 9
Anorexia (Metabolism and nutrition disorders) | 35 | 37
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 5
Dizziness (Nervous system disorders) | 9 | 11
Dysgeusia (Nervous system disorders) | 3 | 10
Headache (Nervous system disorders) | 42 | 49
Neuropathy Peripheral (Nervous system disorders) | 9 | 8
Paraesthesia (Nervous system disorders) | 6 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.